CLINICAL TRIAL: NCT04287621
Title: Registry of Asthma Patients Initiating DUPIXENT® (RAPID)
Brief Title: Registry of Asthma Patients Initiating DUPIXENT®
Acronym: RAPID
Status: Active, not recruiting | Type: Observational
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: R668-AS-1885; EUPAS41963 (Other: HMA-EMA RWD Catalogues)
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Asthma
Keywords: Primary Indication of Asthma
MeSH Terms: conditions — Asthma | interventions — dupilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 156 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: DUPIXENT® — There is no investigational product provided by the study sponsor and no therapeutic intervention regulated by this protocol. As a condition for eligibility, patients are required to initiate DUPIXENT® for asthma, according to the country-specific prescribing information, prescribed by their physician as part of their normal care (ie, not for the purpose of enrolling in the registry). Once patients enter the study, there are no protocol requirements regarding DUPIXENT® or any other treatments.
  Other Names: dupilumab; REGN668; SAR231893

SUMMARY:
The primary objective of the study is to characterize the patients who initiate treatment for asthma with DUPIXENT® in a real-world setting to understand the attributes of treated patients in real life.

This includes characterization of:

* Patient demographics (eg, gender, age, and race)
* Patient baseline characteristics (eg, prior medications and procedures, medical history, asthma history, weight, height)

The secondary objectives of the study are:

* To characterize real-world use patterns of DUPIXENT® for asthma
* To assess the long-term effectiveness of DUPIXENT® in asthma patients in a real-world setting
* To assess effectiveness on comorbid type 2 inflammatory conditions in asthma patients treated with DUPIXENT®
* To collect long-term safety data on study participants in the real-world setting

DETAILED DESCRIPTION:
3-year registry of real-world use of DUPIXENT® for asthma in patients age 12 and over

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to comply with the required clinic visits, study procedures and assessments
* Able to understand and complete study-related questionnaires
* Provide signed informed consent; for patients under the age of 18, both parental (legal guardian) consent and patient assent are required
* Initiating treatment with DUPIXENT® for a primary indication of asthma according to the country-specific prescribing information

Key Exclusion Criteria:

* Patients who have a contraindication to DUPIXENT® according to the country-specific prescribing information
* Treatment with dupilumab within 6 months before the screening visit, or within 6 months of the baseline visit if the screening and baseline occur on the same day
* Any condition that, in the opinion of the investigator, may interfere with patient's ability to participate in the study or personal conditions and circumstances that can predictably prevent the patient from adequately completing the schedule of visits and assessments.

NOTE: Other protocol defined Inclusion/Exclusion criteria apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population comprises adult and adolescent patients (male or female, ≥12 years old), who are initiating treatment with DUPIXENT® for asthma according to the country-specific prescribing information.
Sampling Method: Non-Probability Sample
Enrollment: 718 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2026-05-13 (Estimated); Study Completion 2026-05-13 (Estimated)

PRIMARY OUTCOMES:
Demography | At Baseline
  Including gender, age, race
Baseline Characteristics | At Baseline
  Including prior medications and procedures, medical history, asthma history, weight, height

SECONDARY OUTCOMES:
Baseline Treatment Characteristics | At Baseline
  Including but not limited to treatment dose, frequency, duration and asthma treatment associations.
Incidence of adverse events (AEs) | Baseline up to 3 years
  Including but not limited to: frequency, percentage and exposure-adjusted incidence rate of AEs
Physician Assessment: - Spirometry | Baseline up to 3 years
  Assessment collected as per standard of care. Includes forced expiratory volume in 1 second (FEV1), peak expiratory flow (PEF), forced vital capacity (FVC), forced expiratory flow (FEF) between 25% to 75% of vital capacity (FEF25%-75%), post-bronchodilator FEV1.
Physician Assessment: Fractional exhaled Nitric Oxide (FeNO) | Baseline up to 3 Years
  Assessment collected as per standard of care.
Patient Reported Outcome: Asthma Control Questionnaire, 6-item (ACQ-6) | Baseline up to 3 Years
  Questionnaire assessing the most common asthma symptoms during the previous week, using a 7-point Likert scale (0=fully controlled; 6=severely uncontrolled). Higher score indicates worse asthma control.
Patient Reported Outcome: Mini Asthma Quality of Life Questionnaire (MiniAQLQ) | Baseline up to 3 Years
  Questionnaire answered using a 7-point Likert scale (1=maximum impairment; 7=no impairment). Higher score indicates less impact of asthma on quality of life.
Patient Reported Outcome: Global Patient Assessment | Baseline up to 3 Years
  Assessing patient's symptom severity over the past week and the patient's overall satisfaction with their asthma treatment. Higher scores indicate higher severity of asthma symptoms and lower satisfaction with asthma treatment.
Patient Reported Outcome: Physical Activity Limitation Questionnaire (PALQ) | Baseline up to 3 Years
  Assessing patient's physical activity in their free time. Higher score indicates more health-related quality of life impairment.
Patient Reported Outcome in patients with allergic rhinitis: Allergic Rhinitis Visual Analog Scale (AR-VAS) | Baseline up to 3 Years
  Assessing severity of rhinits symptoms where higher score indicates more bothersome allergic symptoms.
Patient Reported Outcome in patients with allergic rhinitis: Standardized Rhinoconjunctivitis Quality of Life Questionnaire for patients 12 years of age and older (RQLQ[S]+12) | Baseline up to 3 Years
  Health-related quality of life signs and symptoms that are most problematic, as a result of perennial or seasonal allergic rhinitis. RQLQ(S)+12 responses are based on 7-point Likert scale with responses ranging from 0 (not troubled) to 6 (extremely troubled). Higher score indicates more health-related quality of life impairment.
Patient Reported Outcome in patients with chronic (rhino) sinusitis and/or nasal polyps: Sino-Nasal Outcome Test (SNOT-22) | Baseline up to 3 Years
  Questionnaire to assess the impact of chronic rhinosinusitis on quality of life. Lower score represents better health related quality of life.
Patient Reported Outcome in patients with atopic dermatitis: Patient Oriented Eczema Measure (POEM) | Baseline up to 3 Years
  Questionnaire assessing eczema severity with lower score representing impact of lower severity of less severe eczema.
Patient Reported Outcome: Work Productivity and Activity Impairment Questionnaire for asthma (WPAI-asthma) | Baseline up to 3 Years
  Questionnaire to measure impairments in work and activities with higher score indicating greater impairment and less productivity.
Healthcare Utilization: Healthcare Resource Utilization Questionnaire (HCRUQ) | Baseline up to 3 years
  The HCRUQ collects information on unscheduled healthcare resource encounters related to asthma

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (128):
- United States (73):
  - Clinical Research Center of Alabama, LLC, Birmingham, Alabama
  - Arizona Allergy & Immunology Research, Gilbert, Arizona
  - Medical Research of Arizona, a Division of Allergy, Asthma & Immunology Associates, Ltd., Scottsdale, Arizona
  - Children's Hospital of Orange County, Orange, California
  - Riviera Allergy Medical Center, Redondo Beach, California
  - Allergy & Asthma Medical Group and Research, A PC, San Diego, California
  - Bensch Clinical Research, LLC, Stockton, California
  - Allianz Research Institute, Inc., Westminster, California
  - Global Research Solutions, Hollywood, Florida
  - Memorial Healthcare System, Hollywood, Florida
  - Clinical Research Specialists, LLC, Kissimmee, Florida
  - Kratz Allergy & Asthma, Port Richey, Florida
  - GCP, Global Clinical Professionals, St. Petersburg, Florida
  - Allergy & Asthma Diagnostic Treatment Center, Tallahassee, Florida
  - Omni Allergy, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - IACT Health Southeast Lung Associates, Rincon, Georgia
  - Treasure Valley Medical Research, Boise, Idaho
  - Northwestern Medical Group Allergy & Immunology Clinic, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - Asthma and Allergy Center of Chicago, Oak Park, Illinois
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - Velocity Clinical Research, Overland Park, Kansas
  - Dr. Henry J. Kanarek Allergy, Asthma & Immunology, Overland Park, Kansas
  - Family Allergy and Asthma, Louisville, Kentucky
  - Allergy & Asthma Specialists, PSC, Owensboro, Kentucky
  - Schreiber Allergy, Rockville, Maryland
  - Virgo-Carter Pediatrics, Silver Spring, Maryland
  - Chesapeake Clinical Research, Inc., White Marsh, Maryland
  - University of Michigan Allergy Specialty Clinic and Food Allergy Clinic, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Allergy and Asthma Center of Minnesota, Maplewood, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - ENT & Allergy Center of Missouri, Columbia, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - The Clinical Research Center, LLC, St Louis, Missouri
  - Nebraska Medical Research Institute, Inc., Bellevue, Nebraska
  - CHI Health Clinic Pulmonary, Omaha, Nebraska
  - Ocean Allergy & Respiratory Research Center, Brick, New Jersey
  - Atlantic Research Center, LLC, Ocean City, New Jersey
  - A Atat Progressive Pulmonary & Sleep Medicine, Brooklyn, New York
  - New York Allergy and Sinus Centers, Glendale, New York
  - Northwell Health Division of Allergy & Immunology, Great Neck, New York
  - Northwell Health Physician Partners Pulmonary Medicine and Cardiology at Manhasset, Manhasset, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Summit Health, Oakland Gardens, New York
  - RRH Allergy, Immunology & Rheumatology, Rochester, New York
  - Allergy & Asthma Care of LI, Rockville Centre, New York
  - Montefiore Medical Center, The Bronx, New York
  - Allergy Partners of Western North Carolina, Asheville, North Carolina
  - Allergy Partners of the Triangle, Cary, North Carolina
  - UNC Children's Hospital, Chapel Hill, North Carolina
  - Javara Inc. and Tryon Medical Partners, PLLC, Charlotte, North Carolina
  - Airways Clinical Research Center, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Allergy, Asthma and Clinical Research Center, Oklahoma City, Oklahoma
  - Oklahoma Institute of Allergy and Asthma Clinical Research, LLC, Oklahoma City, Oklahoma
  - Portland Research, Happy Valley, Oregon
  - Allergy and Asthma Specialists, P.C., Blue Bell, Pennsylvania
  - Columbo Asthma, Allergy and Immunology, LLC, Bryn Mawr, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Asthma, Nasal Disease & Allergy Research Center of New England, East Providence, Rhode Island
  - National Allergy and Asthma Research, LLC, North Charleston, South Carolina
  - Charleston ENT Associates, LLC, Summerville, South Carolina
  - Precision Research Institute, LLC, Houston, Texas
  - STAAMP Research, LLC, San Antonio, Texas
  - Element Research Group, San Antonio, Texas
  - Tanner Clinic, Layton, Utah
  - Allergy Associates of Utah, Murray, Utah
  - Seattle Allergy & Asthma Research Institute, Seattle, Washington
  - Gundersen Health System, La Crosse, Wisconsin
- Canada (7):
  - The University of British Columbia, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - BLC Clinical Research, Burlington, Ontario
  - Evidence Based Medical Educator Inc., Toronto, Ontario
  - Inspiration Research Limited, Toronto, Ontario
  - Dr. Syeed Anees Medicine Professional Corporation, Windsor, Ontario
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec (IUCPQ) - Universite Laval, Québec
- Sygehus Lillebaelt - Vejle Sygehus - Lungemedicinsk afdeling, Vejle, Denmark
- France (6):
  - Centre Hospitalier du Pays d'Aix - Maladies Respiratoires, Aix-en-Provence
  - CHU de Bordeaux, Bordeaux
  - Centre Hospitalier Universitaire Dijon Bourgogne (CHU Dijon) - Hôpital Francois Mitterrand, Dijon
  - Hôpital de la Croix-Rousse, Lyon
  - Hôpital Nord, Marseille
  - Hopital Jacques Monod, Montivilliers
- Italy (7):
  - Fondazione Salvatore Maugeri, Bari, Apulia
  - Ospedale dei Bambini Vittore Buzzi ASST Fatebenefratelli Sacco, Milan, Lombardy
  - Ospedale Luigi Sacco, PU, ASST Fatebenefratelli Sacco, Milan, Lombardy
  - La Fondazione IRCCS Policlinico "San Matteo", Pavia, Lombardy
  - Istituto Clinico Himanitas, Humanitas Mirasole S.p.a., Rozzano, Lombardy
  - Azienda Sanitaria Locale Salerno, Battipaglia, Salerno
  - Istituto Nazionale di Riposo e Cura per Anziani, Ancona, The Marches
- Japan (12):
  - Hansaki Clinic, Kiyosu-shi, Aichi-ken
  - Hokkaido University Hospital, Kita-ku, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Dokkyo Medical University Hospital, Mibu, Tochigi
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Incorporated Medical Corporation, Shishin Iryokai, Respiratory Care Clinic Tokyo, Chuo-ku, Tokyo
  - Teikyo University Hospital, Itabashi-ku, Tokyo
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
  - Incorporated Medical Corporation, Jinyukai, Jinyu Clinic, Nakano Ku, Tokyo
  - Showa University Hospital, Shinagawa-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - The Fraternity Memorial Hospital, Sumida-ku, Tokyo
- Puerto Rico (6):
  - Agosto Allergy and Immunology, Cayey
  - CardioPulmonary Research CSP, Guaynabo
  - Instituto Pulmonary Diseases Torre Medica San Lucas, Ponce
  - Rafael H Zaragoza - Urdaz, San Juan
  - Fundacion de Investigacion de Diego, San Juan
  - University of Puerto Rico Medical Sciences Campus, San Juan
- Spain (4):
  - Hospital De La Santa Creu I Sant Pau, Barcelona, Catalonia
  - Hospital Universitari Vall d'Hebron, Barcelona, Catalonia
  - Hospital Germans Trias i Pujol, Barcelona, Catalonia
  - Complexo Hospialario Universitario A Coruña, A Coruña, Galicia
- Fysikalisk Medicin, Lidingö, Stockholms Län [se-01], Sweden
- United Kingdom (11):
  - Pennine Acute Hospitals NHS Trust, Manchester, Greater Manchester
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Royal Devon University Healthcare NHS Foundation Trust, Exeter
  - Gartnavel General Hospital, Glasgow
  - St. James Hospital Leeds, Leeds
  - Glenfield General Hospital, Leicester
  - St. Bartholomew's Hospital, London
  - Guy's Hospital, London
  - Wythenshawe Hospital, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Nottingham

REFERENCES:
- [Derived] Gall R, Jain N, Soong W, Settipane RA, Xia C, Zhang Y, Haselkorn T, Jacob-Nara JA, Siddiqui S. Dupilumab-Treated Patients with Asthma in the Real World: The RAPID Global Registry. Adv Ther. 2023 Mar;40(3):1292-1298. doi: 10.1007/s12325-022-02399-5. Epub 2023 Jan 10. PMID 36626107